CLINICAL TRIAL: NCT04129099
Title: A Study of GC022F CAR-T Cell Immunotherapy for Relapsed or Refractory B- ALL
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Collaborators: Gracell Biotechnology Ltd. (Other); Beijing Lu Daopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGC0006
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment group (Experimental): The patients will receive one dose of GC022F. GC022F dosage ranges from 6×10^4 to 1.5×10^5 CAR+T/Kg.
  Interventions: Biological: GC022F

INTERVENTIONS:
Biological: GC022F — GC022F is the CAR-T cell immunotherapy targeted CD19 and CD22. The subjects will receive GC022F as one dose. The dosage ranges from 6×10^4 to 1.5×10^5 CAR+T/Kg.

SUMMARY:
The study is an early, open, single-centered trial. The aim of this study is to evaluate the safety and tolerance of GC022F CAR-T cell immunotherapy in relapsed or refractory B-ALL. The study will include 18 subjects to receive GC022F therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 2-70 years;
2. Eastern cooperative oncology group (ECOG) performance status of 0 to 2;
3. Life expectancy≥12 weeks;
4. CD19 and/or CD22 tumor expression demonstrated in bone marrow or peripheral blood by flow cytometry;
5. Relapsed or refractory B- ALL: a) Refractory B- ALL: MRD≥0.1% or fail to achieve a CR after 2 cycles of a standard induction chemotherapy regimen or one-line/multi-line salvage chemotherapy; b) Relapsed B- ALL: Relapse after remission for the first time in 12 months or relapse after one-line/multi-line salvage chemotherapy; Relapse is defined as MRD≥0.1% or recurrence of primitive cell in peripheral blood or bone marrow(>5%) after remission; c)Relapse after autologous stem cell transplantation or allogeneic hematopoietic stem cell transplantation; Relapse is defined as above; d)Patients with Philadelphia chromosome positive(Ph+) ALL were eligible if they were intolerant to or had failed two lines of tyrosine kinase inhibitor (TKI) therapy, or had t315i mutation.
6. Did not receive hematopoietic stem cell transplantation≤6 months prior to enrollment;
7. Adequate organ function defined as: a) Creatinine clearance (as estimated by Cockcroft Gault) >60 mL/min; b) Serum ALT/AST <2.5 ULN; c) Total bilirubin <1.5 ULN (subjects with Gilbert's syndrome≤3 ULN); d) Cardiac ejection fraction≥50%, no evidence of clinically significant pericardial effusion as determined by an ECHO; e) No clinically significant pleural effusion; f) Baseline oxygen saturation >92% on room air;
8. Females of reproductive age must be in non-lactation period. Females of childbearing potential must have a negative serum or urine pregnancy test. All subjects must use medical-approved-contraception (such as intrauterine device and contraceptive drugs) during the period of trial and in 2 years after cell transfusion therapy; Males should avoid sperm donation;
9. Venous access can be established, peripheral blood mononuclear cells (PBMC) can be collected in researcher's judgement;
10. The subject agrees to and sign informed consent form, willing and able to comply with the planned visit, research, treatment planning, laboratory and other test procedures.

Exclusion Criteria:

1. Isolated extra-medullary disease relapse;
2. Central nervous system leukemia involved CNS-3;
3. Concomitant malignancy other than cured non-melanoma skin cancer or cervical carcinoma in situ or localized prostate cancer or superficial bladder cancer or ductal carcinoma in situ or diagnosis of other malignancy exceeds 5 years without relapse or treatment during the 5 years;
4. Any result of the following virology tests is positive: HIV; HCV; HBsAg; or HBCAb positive with HBV DNA copies positive; TPPA;
5. Live vaccine ≤4 weeks prior to enrollment;
6. For Ph+ ALL, TKI therapy ≤1 weeks prior to enrollment;
7. Presence of ≥ grade 2 acute graft-versus-host disease (GVHD, Glucksberg criteria) or extensive chronic GVHD (Seattle criteria) that require treatment ≤4 weeks prior to enrollment, or during the study period the subject is required to receive anti- GCHD therapy in researcher's judgement;
8. Presence of concomitant disease that require systemic steroids or other immune suppressive therapy during the study period in researcher's judgement;
9. Allogeneic cell therapy (such as donor lymphocyte infusion, DLI) ≤4 weeks prior to enrollment;
10. CNS stereotactic radiotherapy ≤4 weeks prior to enrollment;
11. Toxicities related to previous therapy did not relieved to ≤1 grade, except hematological toxicity and alopecia;
12. Known life-threatening hypersensitivity to cyclophosphamide or fludarabine, or presence of other intolerant conditions, or severe allergic constitution;
13. Patients with active autoimmune disease (e.g., systemic lupus erythematosus, sjogren syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, Hashimoto's thyroiditis, hypothyroidism which can be controlled by thyroid hormone replacement therapy is an exception);
14. For patients that underwent or plan to undergo major surgical operation before CAR-T treatment, surgical operation happened ≤4 weeks prior to enrollment, or did not be fully recovered and clinically stable prior to enrollment, or be anticipated to undergo major surgical operation during the study;
15. Any unstable cardiovascular diseases happened ≤6 months prior to enrollment, including but not limited to, unstable angina, myocardial infarction, heart failure (NYHA grade≥ III grade), severe arrhythmia that require drug interference, cardiac angioplasty/coronary stent implantation/ cardiac bypass surgery ≤6 months prior to enrollment;
16. Presence of central nervous system(CNS) disease or disease history, including epilepsy, cerebral Ischemia/bleeding, dementia, cerebellar disease, any autoimmune diseases that involve CNS;
17. Presence of active infection that require therapy ≤2 weeks prior to apheresis;
18. Any other conditions that researcher think it is inappropriate for the subject to anticipate the trial.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment related Adverse Events, CRS and Neurotoxicity (Safety and tolerability) | 2 years
  Adverse events(AEs) will be collected and graded according to ASTCT consensus(for Cytokine Release Syndrome, CRS and Immune Effector Cell-Associated Neurotoxicity Syndrome, ICANS) and CTCAE v5.0(for AE except CRS/ICANS )

SECONDARY OUTCOMES:
CAR copies and concentration of GC022F in peripheral blood, bone marrow and CSF (amplification and persistence) | 2 years
  GC022F CAR copies and cells in peripheral blood, bone marrow and CSF will be measured by qPCR and FCM in 2 years
Overall response rate of patients who received GC022F infusion (efficacy) | 2 years
  Overall response rate will be estimated as the percents of patients who achieved CR or CRi.
Concentraiton of anti-GC022F antibody after infusion (humoral immune response) | 2 years
  After GC022F infusion, GC022F antibody in peripheral blood will be measured in 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Junfang Yang, Bachelor, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China